CLINICAL TRIAL: NCT00771238
Title: A Pilot Study of Pressure Ulcer Incidence and Change in Existing Pressure Ulcers Comparing Subjects Placed on the TC500 Bed With Standard Beds in the 850-SICU Unit
Brief Title: Pilot Study of Incidence and Change in Existing Pressure Ulcers: TC500 Bed Compared With Standard Beds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hill-Rom (Industry)
Responsible Party: Sponsor
Organization: Baxter Healthcare Corporation (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CR-0095
Record Dates: First submitted 2008-10-10; First posted 2008-10-13 (Estimated); Results first posted 2015-09-28 (Estimated); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Pressure Ulcers
Keywords: pressure ulcers; Therapy mattresses; Incidence of pressure ulcers
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- P500 Mattress (Experimental): The new P500 Low Air Loss mattress will be used to replace the standard mattress for this study arm.
  Interventions: Device: P500 Mattress
- Standard of Care Mattress (No Intervention): Cardiovascular ICU patients that receive standard of care mattress (Total Care Treatment Mattress) and standard pressure ulcer prevention care. All patients had daily skin assessments, as per normal care.

INTERVENTIONS:
Device: P500 Mattress — Study mattress
  Arms: P500 Mattress

SUMMARY:
This pilot study will compare the incidence of pressure ulcers and the change in existing pressure ulcers for patients who are either placed on the new TC500 bed against those placed on the standard ICU bed in the Cardiovascular unit of University of Nebraska Medical Center. Additionally, the cost associated with rental beds will be calculated as well as skin care compliance. Sixty patients will be enrolled (30 per study arm).

DETAILED DESCRIPTION:
This single center convenience sample controlled study will admit all subjects admitted to the Cardiovascular Surgical ICU unit. Subjects can have up to a Stage III pressure ulcer (full thickness ulcer) if they are assessed by the clinical wound team not to require a specialty mattress. This 12 bed ICU will have 6 TC500 beds, and 6 existing Total Care beds. A waiver of consent is requested for initial bed placement, to accommodate normal bed assignments within the facility, however, informed consent will be obtained prior to the collection of data for study purposes. Consented subjects will have primary and secondary diagnoses recorded, as well as pressure ulcer risk assessments, assessment of ventilation / oxygenation support measures, and estimated cardiac condition. They will be followed by daily skin assessments until they reach one of the following study endpoints: 1) discharge from the 850 Cardiovascular SICU unit, 2) have skin breakdown, which in the clinical assessment of the wound team staff would require a specialty bed, 3) expire, 4) withdraw informed consent, or 5) complete the 21 day study period.

Subjects who experience either development of pressure ulcers, or worsening of their skin and/or existing pressure ulcers to the point where a specialty bed is deemed required by the wound team staff will be considered treatment failures, and will be placed on the appropriate mattress identified by the treating staff of the hospital for their admitted condition. If the mattress is a rental therapy mattress, an estimate of the costs to rent this product will be calculated for each patient moving onto a rental mattress.

An assessment of skin care protocol adherence will be performed by the Wound Care team on a daily basis where subjects will be audited as to the percent of prescribed measures implemented.

If subjects require rental therapy beds for pressure ulcer development, the costs associated with this rental will be estimated (# days x average dollar value). These costs will be compared between the rental groups.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects admitted to the 850 Surgical ICU
2. Subjects or their legal reprehensive able to provide written consent for study
3. Subjects must be within the weight limits of the beds (70-500 lbs)
4. Subjects who do not require a specialty bed (subjective assessment by wound team)
5. Subjects are 19 years or older

Exclusion Criteria:

1. Subjects that do not wish to participate
2. Subjects thought to require a different mattress by current clinical bed protocols.
3. Subjects who require pulmonary clearance therapy delivered by a pulmonary mattress.
4. Subjects whose weight is outside of the limits of the bed system.
5. Subjects who have already completed 3 days of this study protocol and are considered completed Subjects.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2008-11; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joyce Black, PhD, RN, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- P500 Mattress: ICU patients placed on a TC500 bed with standard pressure ulcer prevention care
  Total Care P500 Mattress: Study mattress
- Standard Care Arm: ICU patients that receive standard of care mattress (Total Care Treatment Mattress) and standard pressure ulcer prevention care.
Period: Overall Study
Arm/Group | P500 Mattress | Standard Care Arm
Started | 31 | 21
Completed | 31 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: ICU patients in a high acuity Medical / Surgical ICU.
Groups:
- Total: Total of all reporting groups
Arm/Group | P500 Mattress | Standard Care Arm | Total
Number analyzed (Participants) | 31 | 21 | 52
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.1 (11.4) | 54.8 (19.1) | 59.1 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 20 | 9 | 29

OUTCOME MEASURES:

1. Primary Outcome: Indicence of Pressure Ulcers
Description: New pressure ulcers were assessed
Time Frame: at the end of study period (21 days)
Population: Tertiary Care ICU patients
Measure: Number; unit: participants
Arm/Group | P500 Mattress | Standard Care Arm
Number analyzed (Participants) | 31 | 21
participants | 0 | 4

2. Secondary Outcome: Cost of Rental Beds
Description: Cost was measured for Beds/Surfaces that are rented for Wound management / prevention purposes only
Time Frame: End of study
Population: Tertiary Care ICU patients
Measure: Number; unit: US Dollars
Arm/Group | P500 Mattress | Standard Care Arm
Number analyzed (Participants) | 31 | 21
US Dollars | 0 | 4116

ADVERSE EVENTS:
Arm/Group | P500 Mattress | Standard Care Arm
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/21
Other Adverse Events (participants affected / at risk) | 1/31 | 0/21
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | P500 Mattress (N=31) | Standard Care Arm (N=21)
Patient fall out of bed (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Patient was not harmed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No